CLINICAL TRIAL: NCT01703546
Title: Weight Loss & CoMorbidity Resolution With Laparoscopic Adjustable Gastric Band Alone vs. Laparoscopic Adjustable Gastric Band With Gastric Plication
Brief Title: Weight Loss & Comorbidity Resolution With LAGB Alone vs. LAGB With Gastric Plication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Allison Barrett, Principal Investigator, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-277A
Record Dates: First submitted 2012-08-10; First posted 2012-10-10 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Morbid Obesity
Keywords: Morbid Obesity; Weight Loss Surgery; Laparoscopic Adjustable Gastric Band; Laparoscopic Gastric Plication; Imbrication
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LAGB & LGCP (Experimental): All study patients will have the following surgical procedure: Laparoscopic Adjustable Gastric Banding and Gastric Plication (LAGB & LGCP).
  The percent of Excess Body Weight Loss will be monitored at all post op visits.
  Interventions: Procedure: LAGB & LGCP

INTERVENTIONS:
Procedure: LAGB & LGCP — All study patients will have the following surgical procedures: Laparoscopic Adjustable Gastric Band & Laparoscopic Gastric Plication. % Excess Body Weight Loss will be monitored at each post op visit.
  Other Names: Laparoscopic Adjustable Gastric Band & Gastric Plication

SUMMARY:
The purpose of this research study is to evaluate whether combining laparoscopic adjustable gastric band (AKA: lap-band surgery, LAGB) and laparoscopic gastric plication (making tucks in the large curve of the stomach with stitches) to lap-band surgery alone will result in a greater loss of excess weight over time. We anticipate that the average percent of excess body weight loss for study subjects will exceed 29% at 12 months.

DETAILED DESCRIPTION:
Laparoscopic Adjustable Gastric Banding when combined with gastric plication will provide lasting weight loss benefits to patients. We are projecting that the percent of Excess Body Weight Loss (% EWL) will be greater in study subjects when compared with our control group with LAGB alone. Furthermore, it is anticipated that the % EWL in study subjects will be similar to patients who have laparoscopic Roux-En-Y Gastric Bypass.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) > 35
* Meet ASMBS and NIH criteria for Weight Loss Surgery
* ASA Class I - III
* Agree to refrain from any type of weight-loss drug (prescription or OTC)or elective procedure that would affect body weight for the duration of the trial.
* English speaking & comprehension
* Normal mental caliber.

Exclusion Criteria:

* Pregnancy, Liver failure or Kidney failure
* Women of childbearing potential lactating at the time of initial consult or at the time of surgery
* Any condition which precludes compliance with the study
* History or presence of pre-existing autoimmune connective tissue disease or cancer must be evaluated on a case by case basis by the Director of Bariatric Surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2011-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
% Excess Body Weight Loss (%EWL) | 6 months post procedure
  Excess Body Weight is identified pre-operatively and will be monitored during each post operative visit. The percent of Excess Body Weight Loss (%EWL) will be calculated using as a baseline the % Excess Body Weight identified pre-operatively during the subject's initial consult. The change in %EWL at will be calculated at 6 months and 12 months. The %EWL will then be compared to a similar cohort of patients who had the LAGB alone at the same milestones. It is anticipated that study patients' %EWL will be significantly greater.

SECONDARY OUTCOMES:
HgbA1c | 12 months post procedure
  A baseline HgbA1c will be obtained pre-operatively for study patients with a comorbid diagnosis of Type 2 Diabetes. HgbA1C will also be obtained at 6 months and 12 months to evaluate the change from the baseline HgbA1C.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ward, MD, Study Chair — North Shore LIJ Health System, Syosset Hospital, Director of Surgery; Allison Barrett, MD, Principal Investigator — North Shore LIJ Health System Syosset Hospital
Locations (2):
- United States (2):
  - Syosset Hospital - Center for Bariatric Surgical Specialties, 221 Jericho Turnpike, Syosset, New York
  - Syosset Hospital, Center for Bariatric Surgical Specialties, Syosset, New York